CLINICAL TRIAL: NCT04473300
Title: Assessment of Lung Recruitablity of Acute Respiratory Distress Syndrome With SARS-CoV-2 Pneumonia by Electrical Impedance Tomography: a Prospective Observational Study
Brief Title: Assessment of Lung Recruitablity of Acute Respiratory Distress Syndrome With SARS-CoV-2 Pneumonia by Electrical Impedance Tomography
Status: Completed | Type: Observational
Sponsor: Osaka University (Other)
Collaborators: Hospital Rebagliati (Unknown)
Responsible Party: Sponsor
Other Study IDs: ASPEIT
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2020-07

CONDITIONS: Critical Illness; ARDS
Keywords: SARS-CoV-2; electrical impedance tomography; positive end expiratory pressure
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Novel coronavirus (SARS-CoV-2: severe acute respiratory coronavirus 2) pneumonia often develop the acute respiratory distress syndrome (ARDS). Lung protective ventilation strategy consisting of low tidal volume and high positive end-expiratory pressure (PEEP) is recommended. However, it is not clear whether injured lungs from SARS-CoV-2 pneumonia have the same mechanical properties, especially response to PEEP as common ARDS. Therefore, the investigators propose an observational study to analyze respiratory mechanics and lung recruitablity using EIT (electrical impedance tomography) in patients with ARDS due to SARS-CoV-2 pneumonia.

DETAILED DESCRIPTION:
The multi-center prospective observational study will enroll 20 adult ARDS patients under mechanical ventilation from Intensive Care Units (ICUs) in Japan and Peru. Informed consent will be waived due to the nature of observational study. Patients with positive SARS-CoV-2 infection will be included. Prior to initiating the protocol, patients will be sedated deeply with sedatives and/or opioids and paralyzed with a continuous infusion of rocuronium. The distribution of ventilation will be evaluated with EIT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with positive SARS-CoV-2 infection＊
2. Patients with ARDS under mechanical ventilation＊＊
3. Patients ≧ 18 years old

   * Definition of SARS-CoV-2 infection positive: SARS-CoV-2 infection is defined as being positive in RT-PCR (real time reverse transcriptase-polymerase chain reaction) assay using nasal or pharyngeal swab samples.

     * Definition of ARDS is as per the Berlin definition (PaO2/FiO2 ≦ 300 mmHg with PEEP ≧ 5 cmH2O)

Exclusion Criteria:

1. Contraindication for EIT monitoring

   1. Unstable spine or pelvic fractures
   2. Pacemaker, automatic implantable cardioverter defibrillator
   3. Skin lesions between the 4th and 5th ribs where the EIT belt is worn
2. Home mechanical ventilation before inclusion
3. Pregnancy
4. DNR (do-not-resuscitate)
5. Increased intracranial pressure (> 18 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with ARDS due to SARS-CoV-2 pneumonia under mechanical ventilation in intensive care unit.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
The distribution of ventilation | Through study completion (up to 24 hours)
  The distribution of ventilation measured by EIT at PEEP 5 and 15.

SECONDARY OUTCOMES:
Silent spaces | Through study completion (up to 24 hours)
  The changes in dependent and non-dependent silent spaces measured by EIT in PEEP 5 and 15.
Respiratory system compliance | Through study completion (up to 24 hours)
  Respiratory system compliance in PEEP 5 and 15.
Oxygenation | Through study completion (up to 24 hours)
  Oxygenation in PEEP 5 and 15.
Dead space ventilation ratio | Through study completion (up to 24 hours)
  Dead space ventilation ratio in PEEP 5 and 15.

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Yoshida, M.D., Ph.D., Principal Investigator — Osaka University
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No